CLINICAL TRIAL: NCT05424887
Title: A Randomized, Double-blind, Multi-center Phase II Clinical Study to Evaluate the Efficacy and Safety of Two Different Dose Groups of AK3280 in Patients With Idiopathic Pulmonary Fibrosis (IPF) Compared to the Placebo Control Group
Brief Title: A Study to Evaluate the Efficacy and Safety of AK3280 in Patients With Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK3280-2002
Record Dates: First submitted 2022-05-09; First posted 2022-06-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100 mg AK3280 (Experimental): After the 4-week screening period, Eligible subjects will be administered daily 100 mg AK3280 b.i.d. for 24weeks
  Interventions: Drug: AK3280
- 200 mg AK3280 (Experimental): After the 4-week screening period, Eligible subjects will be administered daily 200 mg AK3280 b.i.d. for 24weeks
  Interventions: Drug: AK3280
- placebo (Placebo Comparator): There are placebo controls in each dose cohort to assess the safety profile of the study medication. Subjects will be randomized to receive a placebo simultaneously as those subjects randomized to AK3280.
  Interventions: Drug: Placebo
- Extension Study Cohort (Experimental): The extension study includes a 24-week medication observation period and a 4-week safety follow-up period. Subjects who meet the requirements will enter the extension study after 24 weeks of treatment in the main study. Subjects entering the extension study will continue to orally take AK3280 200 mg for 24 weeks.
  Interventions: Drug: AK3280

INTERVENTIONS:
Drug: AK3280 — Active Substance: AK3280, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: 100 mg AK3280; 200 mg AK3280; Extension Study Cohort
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multi-center phase II clinical study conducted in China to compare the efficacy and safety of two different dose groups of AK3280 in IPF patients compared to the placebo control group.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multi-center phase II clinical study conducted in China to compare the efficacy and safety of two different dose groups of AK3280 in IPF patients compared to the placebo control group. One hundred and five IPF patients who have completed the screening assessment and meet the enrollment requirements will participate in this study and be randomized into 3 treatment groups in a 1:1:1 (35:35:35) ratio: AK3280 200 mg group, AK3280 100 mg group and placebo group; the frequency of medication for each treatment group is twice a day (BID).

This study is divided into a main study and an extension study. The main study includes a 4-week screening period, a 24-week medication observation period, and a 4-week safety follow-up period. The extension study includes a 24-week medication observation period and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who sign the informed consent form before participating in the study.

  2. Patients who understand the importance of complying with the study medication regulations and completing all assessments on time during the entire study process, and agree to strictly abide by the protocol regulations, including the restrictions on concomitant medication during the study process.

  3. Patients aged ≥40 years and ≤80 years at the time of enrollment. 4. Patients diagnosed with IPF within five years before screening (but at least 6 months before the first medication) who meet the standards of the latest American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) 2018 guidelines. The diagnosis of IPF needs to be reconfirmed during the screening assessment.

  5. Patients who have completed the HRCT central review assessment during the screening period or completed the HRCT central assessment within 12 months before screening to confirm the diagnosis of IPF. If the patient is unable to provide pulmonary surgical biopsy pathology, the HRCT image must conform to usual interstitial pneumonia to confirm the diagnosis of IPF. Patients who have undergone pulmonary surgical biopsy as part of the initial diagnosis must submit their pathological slices for central review and assessment.

  6. Patients who cannot tolerate pirfenidone or nintedanib and have received no more than 8 consecutive weeks of regular nintedanib or pirfenidone treatment, or patients who, the investigator considers, are not suitable to receive pirfenidone or nintedanib treatment, or patients who refuse to receive pirfenidone or nintedanib treatment.

  7. Patients with %FVC between 50% and 90% (inclusive) at screening, and hemoglobin-corrected %DLco between 30% and 90% (inclusive).

  8. Patients with relatively stable basic lung function, manifested by a <10% relative difference in FVC values at the screening day and the day before administration. The calculation formula is: (FVC value (L) at screening - FVC value (L) one day before administration) )/(FVC value (L) at screening )× 100% And patients who have no other clinically significant acute exacerbations of IPF determined by the investigators at the screening day and the day before administration.

  9. Patients whose 6MWT distance is ≥100 m without auxiliary support.

Exclusion Criteria:

* 1. Patients suffering from interstitial pneumonia of other known causes.

  2. Patients who plan to undergo lung transplantation within 6 months after screening.

  3. Patients suffering from other clinically significant lung diseases (such as asthma, chronic obstructive pulmonary disease, etc.) in addition to IPF.

  4. Patients suffering from any disease whose life expectancy is less than 12 months other than IPF; or patients requiring long-term medical care, or with limited self-care ability, or the investigator believes that it may affect the patient's participation in the completion of this clinical study, or completion of study-related examinations, or affect safety assessments or efficacy assessments.

  5. Patients who have any evidence or clinically significant adverse physical conditions or abnormal examinations (physical examination, vital signs, ECG or laboratory test abnormalities, etc.) that the investigator believes may affect patient safety or the study endpoint assessments.

  6. Patients with forced expiratory volume in the first second (FEV1)/FVC ratio <0.7 after the use of bronchodilators at screening.

  7. Patients with a positive bronchodilation test, manifested as a ≥ 12% increase in FEV1 and an absolute increase≥200 mL in FEV1 after the use of bronchodilators.

  8. Patients with peripheral capillary blood oxygen saturation (SpO2) at rest <88%.

  9. Patients suffering from any clinically diagnosed connective tissue disease, including but not limited to scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis.

  10. Patients with New York Heart Association (NYHA) heart function classification of Class III-IV.

  11. Renal insufficiency or a history of kidney injury; or creatinine clearance <60 mL/min, calculated using the Cockcroft-Gault formula; or patients with end-stage renal disease requiring dialysis.

  12. Patients with diabetes that is not stably controlled at the time of screening (glycated hemoglobin [HbA1c]> 10%).

  13. Patients hospitalized due to acute exacerbation of IPF within 4 weeks before screening or during the screening period.

  14. Patients currently suffering from malignant tumors or who have been assessed to possibly have malignant tumors (except for localized basal cell carcinoma of the skin or cervical cancer in situ).

  15. Local or systemic infection requiring: i. Hospitalization for ≥24 hours within 4 weeks before screening or during the screening period ii. Use of antibiotics (intravenous, intramuscular injection, oral or inhalation) within 4 weeks before screening or during the screening period

  16. Acute phase of severe lung infection

  17. Active tuberculosis requiring treatment within 12 months before screening

  18. Patients with known immunodeficiency, including but not limited to HIV infection

  19. Patients with acute or chronic hepatitis or patients with known liver cirrhosis

  20. Any of the following circumstances: i. Aspartate aminotransferase (AST) ≥ 2 × upper limit of normal ii. Alanine aminotransferase (ALT) ≥ 2 × upper limit of normal iii. Alkaline phosphatase (ALP) ≥ 2 × upper limit of normal iv. Total bilirubin ≥1.5 × upper limit of normal v. Severe liver damage or end-stage liver disease

  21. Patients who have received any of the following chronic treatment within 4 weeks before randomization or within 5 half-lives (whichever is longer): i. Immunosuppressive or immunomodulatory therapy (such as azathioprine, cyclosporine A, cyclophosphamide, D-penicillamine, interferon, tumor necrosis factor-α antagonist) ii. Cytotoxic drugs (such as colchicine) iii. Pirfenidone iv. Tyrosine kinase inhibitors (such as nintedanib) v. Treatment of pulmonary hypertension (such as endothelin receptor antagonists, phosphodiesterase type-5 inhibitors, riociguat, prostacyclin or prostacyclin analogs) vi. N-acetylcystine vii. Other investigational drug viii. Any unapproved drugs for the treatment of IPF, such as interferon-γ, penicillamine, cyclosporine, and mycophenolate

  22. Patients who have received standardized corticosteroid treatment (oral corticosteroids ≤ 10 mg/day are acceptable) within 4 weeks before screening or during the screening period or who require this treatment during the study period.

  23. Patients who have used P-glycoprotein inhibitors or the substrates of transporters OAT1（Organic Anion Transporter 1）, OAT3（Organic Anion Transporter 3）, OCT2（organic cation transporter 2）, MATE2-K（multidrug and toxin extrusion 2-K）, and MATE1（multidrug and toxin extrusion 1）, with a time interval from the first treatment with the study drug less than five half-lives of the above drugs.

  24. Patients with a history of drinking, drug or chemical abuse, which the investigator judges may harm or affect the patient's complete participation in this study.

  25. Patients with known or suspected peptic ulcers, or patients with palsy, esophageal stenosis, or difficulty swallowing drugs.

  26. Patients who smoked within 3 months before screening or are unwilling to quit smoking during the study period.

  27. Patients whose 12-lead ECG results show QTcF（QT interval corrected using Fridericia's formula） interval > 450 msec in men and QTcF interval> 460 msec in women at screening; or patients with a family or personal history of QT interval prolongation syndrome.

  28. Pregnant or breast-feeding women.

  29. Women and men of childbearing age who are unwilling to use effective contraceptive methods during the study period or at least 3 months after the last administration of the investigational drug.

High-efficiency contraceptive methods for female patients include:

1. Complete abstinence
2. Female sterilization operation (bilateral oophorectomy with or without hysterectomy, total hysterectomy or tubal ligation) at least 6 weeks before receiving study treatment.
3. Male sterilization (at least 6 months before screening). For female patients in the study, the male partners who have undergone vasectomy should be their only partners.
4. Use of oral contraceptives (estrogen and progesterone), and female patients should have used the same contraceptives steadily for at least 3 months before receiving study treatment.
5. Injection or implantation of hormonal contraception or placement of intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception with similar efficacy (failure rate <1%), such as hormonal vaginal ring or transdermal hormonal contraception.

High-efficiency contraceptive methods for male patients include:

1. Vasectomy (a post-vasectomy record proves that there are no sperm in the ejaculation).
2. Having sex with a fertile female who uses the aforementioned high-efficiency contraceptive methods.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
After 24 weeks of continuous medication, the absolute decrease in percentage of the predicted FVC from baseline in the AK3280 treatment group compared to the placebo control group. | Up to 24 weeks
  Change in percentage of the predicted FVC from baseline

SECONDARY OUTCOMES:
Assessment of whether AK3280 prolongs the progression-free survival of IPF subjects compared with the placebo control group within 24 weeks and 48 weeks of medication. | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Progression-free survival is defined as the time from randomization to the first occurrence of any of the following events:
  * The percentage of FVC to the normal expected value (%FVC) achieves an absolute decrease of 10%, or
  * The percentage of DLco to the normal expected value (%DLco) achieves an absolute decrease of 15%, or
  * Non-elective hospitalization due to respiratory events
  * Death
The changes from baseline in %DLco， in the AK3280 treatment group compared to the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  - After hemoglobin correction, the absolute decrease in %DLco
  * DLco will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
The proportion of subjects with a ≥15% absolute decrease in %DLco，in the AK3280 treatment group compared to the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  - After hemoglobin correction, the proportion of subjects with a ≥15% absolute decrease in %DLco
  * DLco will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
The absolute decrease in forced vital capacity (FVC) from baseline ， in the AK3280 treatment group compared to the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  FVC will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
The proportion of patients with a percentage of decrease≥ 10%, ≥ 15% or ≥ 20% in FVC from baseline in each group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  FVC will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
The time to the percentage of decrease in FVC reaching 10% from baseline | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  FVC will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
Within 24 and 48 weeks of medication, the changes from baseline in the 6MWT（six-minute walk test） distance in the AK3280 treatment group compared to the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  The 6MWT distance will be measured at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks after the first administration on D1 respectively.
Within 24 and 48 weeks of medication, the acute exacerbation of IPF subjects - The time from randomization to the first acute exacerbation - The proportion of subjects who experience at least one acute exacerbation | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  A subject needs to meet all 3 criteria below to be judged to have acute exacerbation of IPF:
  * Acute worsening or progression of dyspnea occurs within 1 month (manifested as rapid decline in lung function, worsening of hypoxemia, worsening of irritating dry cough, and worsening of wheezing after exercise, etc.)
  * Chest HRCT（high-resolution computed tomography） shows new diffuse ground glass opacities (GGO) and/or consolidation opacities in both lungs on the background of the original mesh opacities, honeycomb opacities and other manifestations of usual interstitial pneumonia (UIP)
  * Heart failure or fluid overload is ruled out
Within 24 and 48 weeks of medication, the IPF-related mortality, all-cause mortality in IPF subjects | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
The changes from baseline in the SGRQ（Saint George's Respiratory Questionnaire） total score in the AK3280 treatment group compared to the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Saint George's Respiratory Questionnaire Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
  Scores range from 0 to 100, with higher scores indicating more limitations.
The proportion of subjects with changes from baseline in the SGRQ ≥4 points from baseline | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Scores range from 0 to 100, with higher scores indicating more limitations.
Within 24 and 48 weeks of medication, the proportion of patients who have dose adjustments due to AEs in the AK3280 treatment group and the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
Within 24 and 48 weeks of medication, the proportion of subjects who discontinue the medication due to adverse events (AE) in the AK3280 treatment group and the placebo control group | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
Assessment of adverse events | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
Assessment of serious adverse events (SAEs) | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
Number of participants with abnormal vital signs | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Vital signs: include pulse, respiration, body temperature and blood pressure
Number of participants with abnormal Physical examination findings | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Physical examination ： include height, weight, skin, head and neck, mouth, chest, abdomen, lymph nodes, nerves and mind, limbs and other sites
Number of participants with abnormal 12-lead ECG readings | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
Number of participants with abnormal laboratory test results | Main study: Up to 24 weeks; Extended study: Up to 48 weeks
  Laboratory tests：include blood routine examination， blood biochemistry ，urine routine test
Pharmacokinetic endpoint：The maximum plasma drug concentration (Cmax) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Time to peak (Tmax) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Area under the plasma drug concentration-time curve from 0 hour to 12 hours (AUC0-12h) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Area under the plasma drug concentration-time curve extrapolated from 0 hour to infinity (AUC0-∞） of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Oral clearance (CL/F) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Oral volume of distribution (Vd/F) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Terminal half-life (t1/2) of AK3280 and AK3280 M2 | Day 1 and Day 7
Pharmacokinetic endpoint：Accumulation coefficient of AK3280 and AK3280 M2 | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Study Director — Medical Director; Yan Wu, Study Chair — Chief Medical Officer
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No